CLINICAL TRIAL: NCT00331552
Title: Phase I - II Study of Doxil® In Combination With Daily Oral Cyclophosphamide and Herceptin for Patients With HER-2/Neu Positive Disease In Patients With Metastatic Breast Cancer
Brief Title: Doxorubicin Hydrochloride Liposome, Cyclophosphamide, and Trastuzumab in Treating Patients With Stage IV Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hannah Linden, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6139; NCI-2010-00798
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-06

CONDITIONS: HER2-positive Breast Cancer; Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — liposomal doxorubicin; Cyclophosphamide; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): Patients receive oral cyclophosphamide once daily on days 1-28 and pegylated doxorubicin HCl liposome IV over 90 minutes on day 1. Treatment repeats every 4-6 weeks in the absence of disease progression or unacceptable toxicity. Some patients with HER2/neu 3+ disease may also receive trastuzumab IV over 30-90 minutes weekly or every 3 weeks at the discretion of the treating physician.
  Interventions: Drug: pegylated liposomal doxorubicin hydrochloride; Drug: cyclophosphamide; Biological: trastuzumab

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin hydrochloride — Given IV
  Other Names: CAELYX; Dox-SL; DOXIL; doxorubicin hydrochloride liposome; Evacet; LipoDox
Drug: cyclophosphamide — Given orally
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana; Enduxan
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2; monoclonal antibody c-erb-2; monoclonal antibody HER2

SUMMARY:
Drugs used in chemotherapy, such as doxorubicin hydrochloride liposome and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving more than one drug (combination chemotherapy) together with trastuzumab may be a better way to block tumor growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To determine the optimal tolerated dose of Doxil when given in combination with daily oral cyclophosphamide in patients with stage IV breast cancer. (Phase I) II. To determine the efficacy (overall clinical response rate) of the optimal tolerated dose of Doxil when given in combination with daily oral cyclophosphamide and herceptin (for HER2 neu positive patients) in patients with stage IV breast cancer. (Phase II) SECONDARY OBJECTIVES: I. To assess the treatment related toxicity associated with each dose level of this regimen and assess efficacy (overall clinical response rate). (Phase I) II. To assess the safety (treatment related toxicity) of the optimal tolerated dose of Doxil when given in combination with daily oral cyclophosphamide and herceptin (for HER2 neu positive patients) in patients with stage IV breast cancer. (Phase II) III. To assess time to progression and overall survival following treatment with Doxil and daily oral cyclophosphamide and herceptin (for HER2 neu positive patients). (Phase II) IV. To compare the response rate in patients who are heavily pretreated to the response rate in patients who are less heavily pretreated. OUTLINE: This is a phase I, dose-escalation study of pegylated doxorubicin HCl liposome followed by a phase II feasibility study. Patients receive oral cyclophosphamide once daily on days 1-28 and pegylated doxorubicin HCl liposome IV over 90 minutes on day 1. Treatment repeats every 4-6 weeks in the absence of disease progression or unacceptable toxicity. Some patients with HER2/neu 3+ disease may also receive trastuzumab IV over 30-90 minutes weekly or every 3 weeks at the discretion of the treating physician. After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must satisfy either a or b: a) Measurable disease by RECIST criteria; x-rays, scans or physical examinations used for tumor assessment must have been completed within 30 days prior to registration; any non-measurable disease must be assessed within 42 days prior to registration; b) Non-measurable disease only, but MUC-1 antigen level (either CA 27-29 or CEA) is > 2X ULN AND MUC-1 antigen has been documented to have increased by 1.5X prior to registration; x-rays, scans or other tests for assessment of non-measurable disease must have been performed within 42 days prior to registration
* ECOG performance status of =< 2
* ANC >= 1,500 cells/mm^3
* Platelet count >= 100,000 cells/mm^3
* Hemoglobin >= 9.0g/dL
* Creatinine =< 2.5 mg/dL
* In the absence of liver metastases, AST / ALT, alkaline phosphatase and total bilirubin must not exceed 2 x upper limit of normal (i.e., must be =< 2 x upper limit of normal)
* In the presence of liver metastases, AST / ALT, alkaline phosphatase and total bilirubin must not exceed 3 x upper limit of normal (i.e., must be =< 3 x upper limit of normal)
* Have a MUGA scan or 2-d echocardiogram indicating an ejection fraction of >= 50% within 42 days prior to first dose of study drug (the method used at baseline must be used for later monitoring)
* Use an adequate contraceptive method (e.g., abstinence, intrauterine device, barrier device with spermicide or surgical sterilization) during treatment and for three months after completing treatment if of reproductive potential
* Be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study specific screening procedures

Exclusion Criteria:

* Pregnant or lactating women
* History of hypersensitivity reactions attributed to a conventional formulation of doxorubicin HCL or the components of Doxil
* Patients who are HER2-neu positive with cardiac disease that would preclude the use of Doxil or Herceptin are not eligible, including active cardiac disease (i.e., angina pectoris that requires the use of antianginal medication, cardiac arrhythmia requiring medication, severe conduction abnormality, clinically significant valvular disease, cardiomegaly on chest x-ray, ventricular hypertrophy on EKG, uncontrolled hypertension [diastolic greater than 100 mm/Hg or systolic > 200 mm/hg], current use of digitalis or beta blockers for CHF, clinically significant pericardial effusion) and history of cardiac disease (i.e., myocardial infarction documented as a clinical diagnosis or by EKG or any other test, documented congestive heart failure, documented cardiomyopathy, documented arrhythmia or cardiac valvular disease that requires medication or is medically significant)
* Has anthracycline resistant disease defined as a) If anthracycline was given for non-metastatic disease: The cumulative dose of anthracycline exceeds 360 mg/m^ 2 for doxorubicin or 540 mg/m^2 for epirubicin AND the disease-free interval from discontinuation of anthracycline to diagnosis of metastatic disease is < 12 months; b) If anthracycline was given for metastatic disease: The cumulative dose of anthracycline exceeds 360 mg/m^2 for doxorubicin or 540 mg/m^2 for epirubicin AND the patient's disease progressed on anthracycline given as palliative therapy
* Except for the following no other malignancy is allowed: synchronous ipsilateral breast cancer of the same subtype (ER/PR, HER-2/neu), adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer or other stage I or II cancer from which the patient has been disease free for at least 5 years
* Any life-threatening illness other than the malignancy for which they are being treated
* Mental illness
* Have a life expectancy of less than 4 months
* Unwillingness to participate or inability to comply with the protocol for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-02; Primary Completion 2011-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Linden, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyclophosphamide, Doxil 30 mg/m^2, Trastuzumab: Patients receive oral cyclophosphamide once daily on days 1-28 and 30 mg/m^2 pegylated doxorubicin HCl liposome IV over 90 minutes on day 1. Treatment repeats every 4-6 weeks in the absence of disease progression or unacceptable toxicity. Some patients with HER2/neu 3+ disease may also receive trastuzumab IV over 30-90 minutes weekly or every 3 weeks at the discretion of the treating physician.
  pegylated liposomal doxorubicin hydrochloride: Given IV
  cyclophosphamide: Given orally
  trastuzumab: Given IV
- Cyclophosphamide, Doxil 35 mg/m^2, Trastuzumab: Patients receive oral cyclophosphamide once daily on days 1-28 and 35 mg/m^2 pegylated doxorubicin HCl liposome IV over 90 minutes on day 1. Treatment repeats every 4-6 weeks in the absence of disease progression or unacceptable toxicity. Some patients with HER2/neu 3+ disease may also receive trastuzumab IV over 30-90 minutes weekly or every 3 weeks at the discretion of the treating physician.
  pegylated liposomal doxorubicin hydrochloride: Given IV
  cyclophosphamide: Given orally
  trastuzumab: Given IV
Period: Period 1: Doxil 30 mg/m^2 (Phase I)
Arm/Group | Cyclophosphamide, Doxil 30 mg/m^2, Trastuzumab | Cyclophosphamide, Doxil 35 mg/m^2, Trastuzumab
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0
Period: Period 2: Doxil 35 mg/m^2 (Phase I)
Arm/Group | Cyclophosphamide, Doxil 30 mg/m^2, Trastuzumab | Cyclophosphamide, Doxil 35 mg/m^2, Trastuzumab
Started | 0 | 3
Completed | 0 | 3
Not Completed | 0 | 0
Period: Period 3: Phase II
Arm/Group | Cyclophosphamide, Doxil 30 mg/m^2, Trastuzumab | Cyclophosphamide, Doxil 35 mg/m^2, Trastuzumab
Started | 24 | 0
Completed | 22 | 0
Not Completed | 2 | 0
Not completed — Neurological Symptoms | 1 | 0
Not completed — Severe Nausea | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Cyclophosphamide, Doxil, Trastuzumab; Phase II: Cyclophosphamide, Doxil, Trastuzumab: Patients receive oral cyclophosphamide once daily on days 1-28 and pegylated doxorubicin HCl liposome IV over 90 minutes on day 1. Treatment repeats every 4-6 weeks in the absence of disease progression or unacceptable toxicity. Some patients with HER2/neu 3+ disease may also receive trastuzumab IV over 30-90 minutes weekly or every 3 weeks at the discretion of the treating physician.
  pegylated liposomal doxorubicin hydrochloride: Given IV
  cyclophosphamide: Given orally
  trastuzumab: Given IV
- Total: Total of all reporting groups
Arm/Group | Phase I: Cyclophosphamide, Doxil, Trastuzumab | Phase II: Cyclophosphamide, Doxil, Trastuzumab | Total
Number analyzed (Participants) | 6 | 24 | 30
Age, Continuous [Median (Full Range); unit: years] | 49.5 [37 to 72] | 57 [40 to 77] | 56.5 [37 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 23 | 29
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 24 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 4 | 21 | 25
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose and Optimal Tolerated Dose of Pegylated Liposomal Doxorubicin Hydrochloride (Doxil) When Given in Combination With Cyclophosphamide (Phase I)
Description: The dose level in which 2 or more patients develop treatment-related toxicity of grade 3 or higher OR require a dose adjustment following the first course of treatment
Time Frame: Up to 24 weeks
Measure: Number; unit: mg/m^2
Arm/Group | Phase I: Cyclophosphamide, Doxil, Trastuzumab
Number analyzed (Participants) | 6
mg/m^2 | 30

2. Primary Outcome: Efficacy as Assessed by the Overall Clinical Benefit Rate
Description: Count of participants with a clinical benefit (i.e., complete response, partial response, and stable disease).
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Groups:
- Cyclophosphamide, Doxil, Trastuzumab: Patients receive oral cyclophosphamide once daily on days 1-28 and pegylated doxorubicin HCl liposome IV over 90 minutes on day 1. Treatment repeats every 4-6 weeks in the absence of disease progression or unacceptable toxicity. Some patients with HER2/neu 3+ disease may also receive trastuzumab IV over 30-90 minutes weekly or every 3 weeks at the discretion of the treating physician.
  pegylated liposomal doxorubicin hydrochloride: Given IV
  cyclophosphamide: Given orally
  trastuzumab: Given IV
Arm/Group | Cyclophosphamide, Doxil, Trastuzumab
Number analyzed (Participants) | 28
Participants
  Complete response | 0
  Partial response | 6
  Stable disease | 15
  Progressive disease | 7

3. Primary Outcome: Safety as Assessed by Grade 1, 2, 3, 4, Fatal Toxicity, Need for Dose Reduction, Treatment Interruption, or Treatment Discontinuation
Description: Count of participants with grade 1, 2, 3, 4, fatal toxicity, need for dose reduction, treatment interruption, or treatment discontinuation
Time Frame: Periodically during study treatment, up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide, Doxil, Trastuzumab
Number analyzed (Participants) | 30
Participants
  Grade 3 adverse events | 14
  Grade 4 adverse events | 3
  At least one dose held or reduced | 18
  Discontinued due to toxicity | 8

4. Secondary Outcome: Treatment-related Toxicity (Phase I)
Description: Count of phase I participants with treatment related toxicity.
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Doxil 30 mg/m^2: Patients receive oral cyclophosphamide once daily on days 1-28 and 30 mg/m^2 pegylated doxorubicin HCl liposome IV over 90 minutes on day 1. Treatment repeats every 4-6 weeks in the absence of disease progression or unacceptable toxicity. Some patients with HER2/neu 3+ disease may also receive trastuzumab IV over 30-90 minutes weekly or every 3 weeks at the discretion of the treating physician.
  pegylated liposomal doxorubicin hydrochloride: Given IV
  cyclophosphamide: Given orally
  trastuzumab: Given IV
- Doxil 35 mg/m^2: Patients receive oral cyclophosphamide once daily on days 1-28 and 35 mg/m^2 pegylated doxorubicin HCl liposome IV over 90 minutes on day 1. Treatment repeats every 4-6 weeks in the absence of disease progression or unacceptable toxicity. Some patients with HER2/neu 3+ disease may also receive trastuzumab IV over 30-90 minutes weekly or every 3 weeks at the discretion of the treating physician.
  pegylated liposomal doxorubicin hydrochloride: Given IV
  cyclophosphamide: Given orally
  trastuzumab: Given IV
Arm/Group | Doxil 30 mg/m^2 | Doxil 35 mg/m^2
Number analyzed (Participants) | 3 | 3
Participants
  Grade 2 Neutropenia | 0 | 1
  Grade 3 Neutropenia | 0 | 1

5. Secondary Outcome: Time to Progression (Phase II)
Description: Median time to progression. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions or new effusions.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Cyclophosphamide, Doxil, Trastuzumab
Number analyzed (Participants) | 22
months | 6.3 [3.6 to NA] — Upper bound of confidence interval is infinite.

6. Secondary Outcome: Progression-free Survival (Phase II)
Description: Kaplan-Meier estimate assessed at 18 months
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: progression free survival probability
Arm/Group | Phase II: Cyclophosphamide, Doxil, Trastuzumab
Number analyzed (Participants) | 22
progression free survival probability | 0.16 [0.033 to 0.77]

7. Secondary Outcome: Overall Survival (Phase II)
Description: Kaplan-Meier estimate assessed at 18 months
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Phase II: Cyclophosphamide, Doxil, Trastuzumab
Number analyzed (Participants) | 22
survival probability | 0.49 [0.32 to 0.76]

8. Secondary Outcome: Comparison of Clinical Benefit Rate in 2 Subgroups--heavily Pre-treated (1 or More Regimens for Advanced Disease) vs Less Heavily Pre-treated (no Regimens for Advanced Disease) (Phase II)
Description: Count of participants with a clinical benefit (i.e., complete response, partial response, and stable disease).
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Heavily Pre-treated: 1 or more regimens for advanced disease
- Less Heavily Pre-treated: no regimens for advanced disease
Arm/Group | Heavily Pre-treated | Less Heavily Pre-treated
Number analyzed (Participants) | 12 | 10
Participants | 9 | 7

ADVERSE EVENTS:
Arm/Group | Cyclophosphamide, Doxil 30 mg/m^2, Trastuzumab | Cyclophosphamide, Doxil 35 mg/m^2, Trastuzumab
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/3
Other Adverse Events (participants affected / at risk) | 27/27 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclophosphamide, Doxil 30 mg/m^2, Trastuzumab (N=27) | Cyclophosphamide, Doxil 35 mg/m^2, Trastuzumab (N=3)
Leukopenia (Blood and lymphatic system disorders) | 19 | 3
Neutropenia (Infections and infestations) | 18 | 3
Nausea (Gastrointestinal disorders) | 14 | 1
Vomitting (Gastrointestinal disorders) | 3 | 0
Anemia (Blood and lymphatic system disorders) | 8 | 0
Alkaline Phosphatase (Metabolism and nutrition disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 0
Fatigue (General disorders) | 12 | 0
Gastric Reflux (Gastrointestinal disorders) | 2 | 0
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 7 | 1
Mucositis (Gastrointestinal disorders) | 4 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Joint Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 0
Weight Loss (General disorders) | 2 | 1
ALT High (Metabolism and nutrition disorders) | 0 | 1
AST High (Metabolism and nutrition disorders) | 5 | 1
Erythma (Skin and subcutaneous tissue disorders) | 3 | 0
Low Hemoglobin (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 4 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1
Taste Alteration (Metabolism and nutrition disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes